CLINICAL TRIAL: NCT04667572
Title: Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Collagen Cross-Linking in Eyes With Corneal Thinning Conditions
Brief Title: Safety & Effectiveness of the PXL-Platinum 330 System for CXL Using Riboflavin Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cornea Associates of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PXL-330-CAT-2
Record Dates: First submitted 2020-12-02; First posted 2020-12-14 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Keratoconus; Pellucid Marginal Corneal Degeneration; Corneal Degeneration; Corneal Ectasia
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulsed 5mW/cm2 (Experimental): 5mW/cm2, with pulsed mode, 10 seconds on, 10 second off, for 36 minute total treatment time
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution
- Pulsed 8mW/cm2 (Experimental): 8mW/cm2, with pulsed mode, 10 seconds on, 10 second off, for 22 minute and 30 seconds total treatment time
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution

INTERVENTIONS:
Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution — Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea
  Other Names: Corneal Crosslinking

SUMMARY:
Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Collagen Cross-linking in Eyes With Corneal Thinning Conditions

DETAILED DESCRIPTION:
Patients with progressive keratoconus, pellucid marginal degeneration, or at risk for post-refractive corneal ectasia will be recruited and undergo epithelial-on corneal crosslinking with the Peschke PXL-330 system using pulsed, accelerated energy delivery. Patients will undergo monitoring for 1 year, with serial measurements of corneal topography, visual acuity, pachymetry, and visual function.

ELIGIBILITY:
Inclusion Criteria:

* 8 years of age or older
* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits
* Contact Lens Wearers Only:
* Removal of contact lenses (if applicable) for the required period of time prior to the screening refraction: Soft, discontinue 3 days; Soft Extended Wear, discontinue 3 days; Soft Toric, discontinue 3 days; Rigid gas permeable, discontinue 2 Weeks (subjects who cannot function without wearing their contact lenses, may forgo discontinuation of contact lenses)

And one or more of the following:

* Presence of central or inferior steepening.
* Axial topography consistent with keratoconus, post-surgical ectasia, or pellucid marginal degeneration
* Presence of one or more findings associated with keratoconus or pellucid marginal degeneration, such as: Fleischer ring, Vogt's striae, Decentered corneal apex, Munson's sign, Rizzutti's sign, Apical Corneal scarring consistent with Bowman's breaks, Scissoring of the retinoscopic reflex, Crab-claw appearance on topography
* Steepest keratometry (Kmax) value ≥ 47.20 D
* I-S keratometry difference > 1.5 D on the Pentacam/Orbscan map or topography map
* Posterior corneal elevation >16 microns
* Thinnest corneal point >300 microns

Exclusion Criteria:

* Eyes classified as either normal or atypical normal on the severity grading scheme.
* Corneal thickness < 300 microns measured by ultrasonic pachymetry or pentacam.
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example: History of or active corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, etc.) Clinically significant corneal scarring in the CXL treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross-linking procedure.
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests.
* Patients with a current condition that, in the physician's opinion, would interfere with or prolong epithelial healing

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
K-Max | 12 Months
  Change in K-Max measured by corneal topography, compared to baseline
K-Mean | 12 Months
  Change in K-Mean measured by corneal topography, compared to baseline

SECONDARY OUTCOMES:
Uncorrected Visual Acuity | 12 Months
  Change in uncorrected corrected visual acuity using snellen measurements, compared to baseline
Best Corrected Visual Acuity | 12 Months
  Change in best corrected visual acuity using snellen measurements, compared to baseline
Central Pachymetry | 12 Months
  Change in central pachymetry, measured by Pentacam compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cornea Associates of Texas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No